CLINICAL TRIAL: NCT06947278
Title: Preoperative Study of the Correlation Between BDNF-TrkB Signaling Pathway Expression Levels in Cerebrospinal Fluid and Blood and Postpartum Depression
Status: Completed | Type: Observational
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Other Study IDs: KY-20240701001-02
Record Dates: First submitted 2025-04-12; First posted 2025-04-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Depression (PPD)
Keywords: prospective observational studies;; Postpartum Depression(PPD); brain-derived neurotrophic factor (BDNF); Edinburgh postnatal depression scale (EPDS); Hamilton depression scale (HAMD-21)
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cerebrospinal fluid and blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This single-center prospective observational study will screen 200 parturients with combined lumbo-epidural anesthesia in the First People's Hospital of Lianyungang City, collect the basic information of the patients, as well as the scores of PSQI, STAI, NRS, SSRS and other scales one day before surgery, and analyze their effects on the expression level of BDNF. On the day of surgery, 10mL of peripheral arterial blood and 3 mL of cerebrospinal fluid were collected, and the expression levels of BDNF-TrkB signaling pathway (ProBDNF, mBDNF, TrkB, P-CREB and ALB) were measured, respectively. The patient's EPDS and HAMD-21 scores were evaluated and collected by a professional psychologist at 1 day before surgery, 7 days after surgery, and 42 days after surgery, and the correlation between BDNF expression level and the occurrence of postpartum depression was statistically analyzed, as well as which in cerebrospinal fluid and blood was more sensitive for predicting postpartum depression.

DETAILED DESCRIPTION:
On the day before delivery, the anterior will explain the purpose of the test to the pregnant woman during the preoperative follow-up, and collect the basic information of the pregnant woman (age, gender, BMI, gestational age, education level, economic status) and the scores of PSQI, STAI, NRS, SSRS and other scales after obtaining the consent of the pregnant woman and signing the informed consent form. On the day of surgery, an anesthesiologist with more than five years of work experience collected 3ml of peripheral blood and 0.5ml of cerebrospinal fluid before anesthesia administration, and measured the expression level of BDNF-TrkB signaling pathway (ProBDNF, mBDN). 1 day before delivery, 7 days and 42 days postpartum were evaluated by a psychologist with more than five years of work experience and collected the patient's EPDS and HAMD-21 scores, the data collection for 1 day before delivery was carried out in the ward, and the follow-up at 7 days and 42 days after delivery was carried out through WeChat questionnaire link and telephone, if no response was received, WeChat contact and phone reminder would be made again after 1 and 2 weeks, if there was still no response, the subject was considered to have missed the postoperative follow-up time and was regarded as missing follow-up, Statistical analysis was performed to analyze the correlation between BDNF expression level and the occurrence of postpartum depression, and which was higher in cerebrospinal fluid and blood for predicting postpartum depression. If the EPDS score is ≥ 9 points, the HAMD-21 score is ≥ 9 points, and the mother has no suicidal tendencies, psychologists will provide psychological support treatment until the score returns to normal; If the woman is suicidal, it is recommended that the patient and her family have agreed to be admitted to the hospital. Subject files will be kept for up to 5 years after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the indications for cesarean section and have no contraindications to neuraxial anesthesia;
2. 20 years old≤ age ≤ 35 years old;
3. 37≤ gestational age< 42;
4. American Society of Anesthesiologists (ASA) grade II~III;
5. singleton pregnancy;
6. Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Unable to understand the content of the questionnaire correctly;
2. a clear history of mental illness, depression, cognitive impairment and other diseases;
3. Patients who have been taking sedative, analgesic and psychotropic drugs for a long time;
4. Those who have recently used glucocorticoids or immunosuppressants;
5. Those who are allergic to or have contraindications to any of the drugs used in this study;
6. Serious pregnancy complications, such as preeclampsia, placental hyperplasia, etc.;
7. Participated in other clinical studies within the last 3 months.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing elective cesarean section under combined lumbar-rigid anesthesia in the First People's Hospital of Lianyungang City
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-16 (Actual); Study Completion 2025-11-16 (Actual)

PRIMARY OUTCOMES:
Correlation between the expression level of BDNF-TrkB signaling pathway (mBDNF, proBDNF) in cerebrospinal fluid and blood and postpartum depression; | Blood and cerebrospinal fluid samples were collected before anesthesia administration on the day of surgery, placed in a -80 degree Celsius freezer, and mBDNF and proBDNF concentrations were measured within 3 months after sample collection.

SECONDARY OUTCOMES:
Comparison of the sensitivity of cerebrospinal fluid and blood levels of BDNF in predicting postpartum depression; | Blood and cerebrospinal fluid samples were collected before anesthesia administration on the day of surgery, placed in a -80 degree Celsius freezer, and BDNF concentrations were measured within 3 months after sample collection.
The correlation between BDNF (mBDNF, proBDNF) concentrations in cerebrospinal fluid and blood. | Blood and cerebrospinal fluid samples were collected before anesthesia administration on the day of surgery, placed in a -80 degree Celsius freezer, and albumin concentrations were measured within 3 months after sample collection.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Lianyungang Hospital of Xuzhou Medical University, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No